CLINICAL TRIAL: NCT02164656
Title: Mindfulness Training for Smokers Online Feasibility Study
Acronym: MTS3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0247; K23DA022471 (NIH)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Cigarette Smoking; Mindfulness
MeSH Terms: conditions — Cigarette Smoking | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mindfulness training (Experimental): 8 week course in mindfulness for smokers
  Interventions: Behavioral: mindfulness for smokers

INTERVENTIONS:
Behavioral: mindfulness for smokers

SUMMARY:
The Mindfulness Training for Smokers Online Feasibility Study is a pilot study designed to test Mindfulness Training for Smokers in an Internet format with phone counseling.

DETAILED DESCRIPTION:
The MTS Online Feasibility Study is funded for through a five-year K23 NIH training grant awarded to Dr. James Davis, the Principal Investigator on this protocol. The study enrollment goal is N=50 adult smokers. MTS Online is an Internet-based smoking cessation intervention that provides access to video material and instructional support for 8 mindfulness classes over a 6-week period. The MTS Online Feasibility Study aims to explore the feasibility of an Internet-based version of MTS, specifically looking at issues of on-line participation and Internet site use, adherence to instructed mindfulness practice regimen, and overall acceptability of MTS Online to a smoking population.

Participants will be recruited for MTS Online through existing recruitment mechanisms already in place for MTS. Specifically, participants who decline or are excluded from the MTS Study due solely to scheduling conflicts will be offered participation in MTS Online. All other inclusion/exclusion criteria are identical to the MTS study and discussed below.

After a decline or exclusion from the MTS Study due to scheduling and no other reason, research assistant will ask the caller if they would like the phone number for the Wisconsin Tobacco Quit Line and will ask the caller if they would like to hear about an online version of the MTS program. If the participant says they are interested, the RA will read a description of the online program and phone screening through the MTS Online Phone Screening Script. This script includes all inclusion and exclusion criteria found in the MTS Study, with the exception of the question on whether the caller can attend all the class meetings. If at the end of the phone script, the caller decides that they would like to come in for an Orientation Meeting, they will be sent an email providing instructions for scheduling their Orientation Meeting.

During the Orientation Meeting/Study Visit 1 MTS staff will provide a general description of the study and review the study consent form. If potential participants choose to join the study they will sign the consent form. After signing consent potential participants will be provided instruction on the use of nicotine patches, smoking calendars and will be provided with intervention materials. Research Assistants will assist participants as they log onto the MTS Online website and create a unique user ID. This ID will be used for all MTS Online features including communicating through the online forum and viewing instructional videos. Potential participants will be given a course schedule with a "class time" for their first class. After this, participants will fill out a Scan Form Questionnaire and proceed to collection of clinical measurements.

Intervention/Study Sign Up: During the Orientation potential participants will be provided with instructions on how to sign up for the intervention and study. This will include the following steps that must be completed through the individual's own Internet access (i.e. not completed at UW-CTRI).

1. Sign on to the MTS Online Forum using the username and password provided during the orientation.
2. Respond to the question "Do you want to join the MTS Online Study?" with the answer "Yes." Participants will be asked to review Class 1 in the MTS Instructional Video and MTS Manual before or during the time scheduled for Class 1. After this time, participants will be asked begin using various mindfulness practices and answer some questions provided by their instructor on how the practices went. This takes place primarily on the MTS Forum where other class participants can benefit from the interaction. Participants will, however, also have access to the instructors email address for private interactions.

Nicotine Replacement Therapy (NRT): All participants will receive two weeks of nicotine patches to start on their Quit Day. Patches will be provided by the MTS Study and mailed directly to PO Box or home address provided by participants approximately 10 days prior to their Quit Day (to assure ample time for delivery). Patch dosing for all participants will be as follows:

14 mg patches for participants who smoke 10 or fewer cigarettes per day 21 mg patches for participants who smoke over 10 cigarettes per day

MTS Online: Participants will have access to 8 classes over a 6-week period through the MTS Online website - www.sittoquit.org. The first 5 classes include instruction through the MTS Instructional Video and MTS Manual. The last 3 classes are provided through materials in the MTS Manual alone. The MTS website contains forum designed specifically for the MTS Online Participants. On this forum, MTS Online Feasibility Study participants can discuss topics related to smoking and mindfulness in discussion groups moderated by MTS mindfulness instructors. Participants will also be provided with the MTS Audio-CD that contains guided mindfulness exercises.

MTS Online Classes: MTS Online classes are provided through the MTS Instructional Video and MTS Manual. The classes provide instruction in mindfulness mediation, mindful walking, mindful eating, and other mindfulness exercises. MTS Online classes provide instruction on how to use mindfulness skills to manage relapse challenges such as smoking triggers, craving, withdrawal symptoms, strong emotions, and stressful situations. The forum serves as a quit smoking support group and provides a place for participants to learn from one another's challenges and through the guidance of a mindfulness instructor. MTS Online classes are available through the MTS Online website. The classes will follow a regular schedule in which participants are to have watched the video material by a certain date (see course schedule above). Following this time, a forum discussion will begin on the website, moderated by the MTS Online mindfulness instructor.

MTS Online Quit Day: Guidelines will be provided to participants for conducting their own personal Quit Day. Participants are encouraged to set aside additional time for mindfulness practice during their Quit Day. Online forum discussion will also take place on the Quit Day. Nicotine patches will be started on the Quit Day and will be continued for 2 weeks.

MTS Online Instructors: Five instructors will moderate various waves of MTS Online. These five include the three instructors who have been trained to teach the Mindfulness Training for Smokers Intervention (see Key Personnel). In addition, the study PI, Dr. James Davis, and a graduate student working on the project, Simon Goldberg, will co-facilitate the early waves. All five MTS Online instructors have completed UW IRB modules provided for Research on Human Subjects. The three MTS instructors have been teaching the MTS course for the last 12 months. MTS Instructors have education the equivalent of a BA/BS or higher and have 2 or more years experience teaching meditation and mindfulness practices. MTS Instructors have completed the MTS Instructor Training Course provided over a weekend. MTS Instructor Training includes standard methods normally provided at CTRI including HIPPA training and UW-IRB training for individuals involved in research on human subjects. Instructor Training also includes instruction on how to conduct MTS including training to familiarize instructors with the MTS Instructional Video, MTS Audio CD and MTS Manual. The list of Key Personnel on the IRB protocol will be updated as new instructors are trained.

MTS Instructional Video: The MTS Instructional Video is a 2-hour DVD course with interviews provided by multiple nationally recognized experts on mindfulness and smoking addiction. It describes how to apply mindfulness to overcome obstacles in smoking addiction. The video is divided into five chapters, one chapter for each class prior to the Quit Day. Most chapters are 15- 20 minutes long. The chapters will provide the primary course material for MTS Online. Participants will be instructed to watch portions of the video on a pre-specified schedule (see above) and participate in forum discussion on topics addressed in the video.

MTS Manual: The MTS Manual contains organizational materials, conceptual information and class exercises. It follows the format of the MTS Video but expands on the information. The manual is intended to reinforce and expand participants understanding of how to use mindfulness to quit smoking.

MTS Website: The MTS website is available through the URL: www.sittoquit.org. The MTS website contains a 2-minute video on the homepage that provides information on the study and intervention. MTS Online participants will be able to gain access to other parts of the web site by use of a unique login name and password created during the Orientation Meeting/Study Visit 1. The MTS website contains a meeting calendar, the MTS Instructional Video, the MTS Manual and the MTS Online Forum specially designed so that participants in the MTS Online Feasibility Study can interact with MTS Instructors and other participants. An additional forum exists for non-Online participants (i.e. participants in the non-online MTS study). The website is maintained through University of Wisconsin information technology services. Activity on the web site will be monitored by the PI and by a UW CTRI IT specialist.

Daily Meditation/MTS Audio CD: MTS Online participants will be asked to meditate each day with the MTS Audio CD starting after their first mindfulness class and continuing until 1 month after their Quit Day, although participants will be encouraged to practice meditation indefinitely. The MTS Audio-CD contains a 15-minute and a 30-minute guided meditation practice. The CD was made by Dr. James Davis and provides instructions for mindfulness meditation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years or over
2. Participants must express "high" motivation to quit smoking
3. Participants must smoke 5 or more cigarettes per day

Exclusion Criteria:

1. Self report of alcohol use of 4 drinks or more a night on 4 or more nights per week.
2. Self report of using chewing tobacco, snuff or cigars in the last week
3. Severe depression or suicidality as assessed via the Patient Health Questionnaire (see section below for details)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Biochemical Abstinence Testing | 4 and 24 week post quit attempt
  Carbon Monoxide Breath Test (CO): CO is expired in detectable levels for up to 48 hours after smoking and can provide verification of tobacco use or abstinence. CO breath test is provided via a calibrated CO breath monitor. Per standard CTRI protocol, a cut-off value of less than 7 ppm will be employed to verify abstinence. Breath testing will be conducted at baseline, at 4 weeks post-quit and at 24 weeks post-quit.

SECONDARY OUTCOMES:
Five Factor Mindfulness Questionnaire | baseline, 4 and 24 months post quit
  Five Factor Mindfulness Questionnaire
Depression, Anxiety and Stress Scale | 0, 4 and 24 months
  Depression, Anxiety and Stress Scale
Experiential Avoidance Scale | 0, 4, 24 months
  Experiential Avoidance Scale
Perceived Stress Scale | 0, 4, 24 months
  Perceived Stress Scale
MTS Online Course Evaluation | 4 months post quit

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin School of Medicine, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Davis JM, Manley AR, Goldberg SB, Stankevitz KA, Smith SS. Mindfulness training for smokers via web-based video instruction with phone support: a prospective observational study. BMC Complement Altern Med. 2015 Mar 29;15:95. doi: 10.1186/s12906-015-0618-3. PMID 25886752